CLINICAL TRIAL: NCT02169674
Title: Sustaining Protection Against Hepatitis B From Infancy to Adulthood: Assessing the Case for a Booster Dose in Adolescence
Brief Title: Hepatitis B Booster Study in Adolescence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Immunization Research Network (Network); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, David Scheifele, Clinical Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H13-00049
Record Dates: First submitted 2014-06-11; First posted 2014-06-23 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Vaccine; Immunogenicity
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: A prospective, single-center, parallel group study of residual HBV seroprotection rates and the capacity of seronegative individuals to respond to a challenge dose of HBV vaccine.
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10-11 Year-olds (Active Comparator): Recombinant hepatitis B virus vaccine (EngerixB, GlaxoSmithKline Vaccines)
  Interventions: Biological: EngerixB, GlaxoSmithKline Vaccines
- 15-16 Year-olds (Active Comparator): Recombinant hepatitis B virus vaccine (EngerixB, GlaxoSmithKline Vaccines)
  Interventions: Biological: EngerixB, GlaxoSmithKline Vaccines

INTERVENTIONS:
Biological: EngerixB, GlaxoSmithKline Vaccines

SUMMARY:
This study looks at protection in 10-11 and 15-16 year olds, immunized as infants with Hepatitis B (HB) vaccine to see if they still have residual protection against Hepatitis B disease. Adolescents will be invited to have a blood test and those without a minimal level of protection (antibody titer) will be offered a "test" vaccination to see if they still have capacity to recall an immune response. About one month later they will get another blood test to see if a booster response occurred. A few participants will have lost protection (no booster response) and will be offered a second HB vaccination to restore protection. Results of this study could influence the way in which children in British Columbia (BC) are immunized against HB disease.

DETAILED DESCRIPTION:
Purpose:

The purpose of the study is to assess whether or not individuals immunized as infants with Hepatitis B vaccine have residual immunity in their pre-adolescent and adolescent years. Two age groups (10, 11 year olds and 15, 16 year olds) will be invited to have blood taken to measure their level of protection (antibody titer). Those without a minimum protective titer will be offered a Hepatitis B "test" vaccination to determine if they still have the capacity to recall an immune response (ie immune memory), as a second line of protection against infection. A second blood sample will be obtained to determine if a booster response occurred (immune memory persists, protection intact) or not. The study vaccine will be a pediatric dose of HB vaccine (EngerixB) made by GlaxoSmithKline Canada (10mcg), a licensed product used in the public immunization program in British Columbia (BC) currently.

Hypothesis:

The hypothesis being tested is that protection has been lost in a sufficient proportion of 15-16 year olds to warrant consideration of a pre-adolescent HB booster, modeled by the 10-11 year olds whose protection is expected to be uniformly reinforceable.

Justification:

This will be the first Canadian study of the duration of the HB immune memory after infant immunization. According to a systematic review of 46 studies, evidence of progressive loss of immune memory and protection decades after infant HB vaccination is clear. Provinces in Canada recently took a leap of faith in dropping their adolescent HB immunization programs, assuming that HB protection from infancy will be life-long. This project investigates residual HB immunity 10 and 15 years after infant vaccination and evaluates a prototype booster program to provide health officials with timely, strategic information for maintaining optimal, informed HB disease control.

Research Methods:

The study will be conducted in BC which has used a consistent infant HB dosing schedule throughout. Eligible participants will be healthy 10-11 or 15-16 year olds. After obtaining informed consent/assent, a blood sample (8 ml) will be obtained to measure serum anti-HBs (anti-HB surface antigen) titer. Participants with a titer ≥10 IU/L will be informed of their ongoing protection and will exit the study. Those with a titer of ≤10 IU/L will be invited to return for a second visit for an HB challenge immunization. Participants will be asked to return 28 days post-vaccination for another blood test. Those who developed a booster response will be informed that they are immune and will exit the study. Those who do not boost will be invited to return for an additional (remedial) HB vaccination with a final titer check available to confirm restoration of protection. Tests will be carried out at BC Center for Disease Control's Hepatitis Laboratory. Booster responses are expected to be strong (titers >100 IU/L). Samples with post-booster titers 10-99 IU/L may be retested to assess antibody avidity to distinguish between primary and secondary type responses.

Data will be assembled by the study center team. Electronic case report forms will capture case and laboratory information, using a commercial platform.

Statistical Analysis Plan The baseline blood test will identify participants with residual anti-HBs titers above or below the minimum protective threshold of 10 IU/L. Based on the meta-analysis of studies involving 10 or 15 years of follow-up after infant immunization, the investigators project that about 30% of younger and 60% of older participants will have titers <10 IU/L. The booster challenge will identify those who are able to mount an anamnestic/recall response (titer ≥100 IU/L), a possible primary response (titer 10-99 IU/L, low avidity) or no response (titers <10 IU/L). The investigators project that 25-30% of older booster recipients will not have an anamnestic response, representing 15-20% overall of that study population. To detect a susceptibility rate of 15% with a precision of ± 0.05 and 95% confidence intervals, it will be necessary to screen 220 individuals, allowing for a 10% drop-out rate. Among younger booster recipients, the investigators project that 10% will not have an anamnestic response, representing an overall susceptibility rate of ~3%. For a precision ± 0.03 and 95% confidence intervals, the number of younger subjects to be screened will be 140, allowing for a 10% drop-out rate.

Multivariable analysis will be undertaken to identify factors associated with loss of detectable protection, such as age at final dose, interval since vaccination, gender etc. The apparent rate of decline in titers between 10 and 16 years of age will be calculated.

Mathematical modelling and economic analysis of immunization program options will be included to aid subsequent decision-making by health authorities. Among the options to be modelled are no intervention (relying on herd immunity of adjacent age groups) and a single booster dose at age 10-11years (grade 6 in BC, the locus of the cancelled adolescent HB vaccination program).

ELIGIBILITY:
Inclusion Criteria:

* Age 10-11 or 15-16 years
* Written informed assent provided by 10-11 year old participants and consent by their parent or legal guardian OR written informed consent provided by a 15-16 year old participant.
* Subjects whom the investigator believes can and will comply with the requirements of the protocol.
* General good health
* Immunized in BC on the regular schedule with hepatitis B vaccine at approximately 2, 4, 6 months of age, based on an available immunization record.

Exclusion Criteria:

* Hepatitis B vaccination regimen for infants born to a mother with hepatitis B infection (e.g. doses at birth and ages 1 and 6 months, with or without HB immune globulin at birth).
* Receipt of any additional dose(s) of hepatitis B vaccine beyond infancy.
* Systemic hypersensitivity to hepatitis B vaccine or severe reaction to any previous dose of hepatitis B vaccine.
* Receipt of blood or blood product within 3 months prior to Visit 1.
* Immune compromise resulting from disease or immunosuppressive systemic medication use within 3 months prior to Visit 1.
* Chronic health condition requiring ongoing medical supervision e.g. cystic fibrosis.
* Incapacity to provide fully informed assent, resulting from cognitive impairment.
* Inadequate participant or parental (when the parent will provide consent) fluency in English to provide fully informed consent.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 359 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Scheifele, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vaccine Evaluation Center (University of BC at Children's Hospital), Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Pinto M, Dawar M, Krajden M, Naus M, Scheifele DW. Will Infant Hepatitis B Vaccination Protect Into Adulthood?: Extended Canadian Experience After a 2-, 4- and 6-month Immunization Schedule. Pediatr Infect Dis J. 2017 Jun;36(6):609-615. doi: 10.1097/INF.0000000000001543. PMID 28134742
- See also: click here for information on the trial — http://www.vec.med.ubc.ca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening for eligibility will be part of volunteer identification, with confirmation of eligibility to follow at the first in-person visit. A component of volunteer screening will be initiating a review of individual HBV immunization records.
Pre-assignment Details: Initially, 359 volunteers who met inclusion criteria where recruited, of whom 6 were deemed ineligible due to late disclosure of neonatal HBV vaccination (n=3), ineligible medical condition (n=2) or additional doses of HBV vaccine (n=1). Three early consent withdrawals resulted in 350 participants who underwent baseline testing.
Groups:
- 10-11 Year-olds; 15-16 Year-olds: Single challenge dose of HBV vaccine (10 mcg, Engerix B, GSK)
Period: Overall Study
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Started | 137 | 213
Completed | 105 | 135
Not Completed | 32 | 78
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Seroprotected | 30 | 76
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10-11 Year-olds | 15-16 Year-olds | Total
Number analyzed (Participants) | 137 | 213 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 137 | 213 | 350
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (0.50) | 16.0 (0.18) | 13.9 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 87 | 156
  Male | 68 | 126 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 78 | 99 | 177
  Chinese | 18 | 55 | 73
  South Asian | 6 | 6 | 12
  Mixed | 29 | 35 | 64
  Other | 6 | 18 | 24
Region of Enrollment [Number; unit: participants]
  Canada | 137 | 213 | 350

OUTCOME MEASURES:

1. Primary Outcome: Serum Anti-HBs Concentration 12 IU/L or Greater
Description: The primary outcome measure is the number of participants who have residual HB immunity 10 or 15 years after infant HB immunization, defined by a persistent anti-HBs titer >12 IU/L.
Time Frame: 10 or more years after infant HB immunization
Measure: Count of Participants; unit: Participants
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Number analyzed (Participants) | 137 | 213
Participants | 30 | 76

2. Primary Outcome: Recollection of Anti-HBs Titer >12 IU/L After Booster
Description: The primary outcome measure is the number of participants who have capacity to recall anti-HBs titer >12 IU/L after HB booster vaccination.
Time Frame: 28 days after HB booster
Measure: Count of Participants; unit: Participants
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Number analyzed (Participants) | 105 | 135
Participants | 102 | 123

3. Other Pre Specified Outcome: Geometric Mean Concentration of Anti-HBs
Description: The geometric mean concentration of anti-HBs antibodies before and after booster vaccination, in both age groups
Time Frame: Before and after booster immunization
Population: Post challenge number analyzed are those nonseroprotected at baseline minus two withdrawals in the 10-11 year-old group and one withdrawal and one loss to follow-up in the 15-16 year-old group.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Number analyzed (Participants) | 137 | 213
mIU/ml
  Before booster | 4.2 [3.38 to 5.22] | 7.98 [6.37 to 9.99]
  After booster: number analyzed (Participants) | 105 | 135
  After booster | 590.6 [473 to 737] | 319.3 [229 to 445]

4. Other Pre Specified Outcome: Anti-HBc (Hepatitis B Core Antigen) Antibody
Description: The number of baseline serum samples that contain anti-HBc antibodies, as a function of time since immunization
Time Frame: Baseline sample
Measure: Count of Participants; unit: Participants
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Number analyzed (Participants) | 137 | 213
Participants | 0 | 0

5. Other Pre Specified Outcome: HBs Antigenemia
Description: The number of baseline serum samples that contain HBs antigen, as a function of time since immunization.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Number analyzed (Participants) | 137 | 213
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | 10-11 Year-olds | 15-16 Year-olds
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/213
Other Adverse Events (participants affected / at risk) | 0/137 | 0/213

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No